CLINICAL TRIAL: NCT05890482
Title: Islamic Trauma Healing: A Scalable, Community-based Program for War and Refugee Trauma
Brief Title: A Scalable, Community-based Program for War and Refugee Trauma
Acronym: ITH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Washington (Other)
Collaborators: Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Lori Zoellner, Professor: Psychology, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00015447; R2HC #70165 (Other Grant/Funding Number: Enhancing Learning & Research for Humanitarian Assistance)
Record Dates: First submitted 2023-02-20; First posted 2023-06-06 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-05

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Islamic Trauma Healing (ITH) (Experimental): A lay-led, six-session group intervention that combines empirically supported exposure-based and cognitive restructuring techniques with Islamic principles.
  Interventions: Behavioral: Islamic Trauma Healing
- Wait List/Delayed (ITH) (Other): Six week waitlist condition and then crossed-over to six weeks of the ITH intervention
  Interventions: Behavioral: Islamic Trauma Healing

INTERVENTIONS:
Behavioral: Islamic Trauma Healing — Manualized, lay-led psychosocial intervention

SUMMARY:
In low and middle-income countries, access to state-of-the-art mental health care is often limited. Islamic Trauma Healing (ITH) is a manualized mosque-based, lay-led group intervention aimed at healing the individual and communal mental wounds of war and refugee trauma. The investigators will execute a hybrid effectiveness-implementation randomized controlled trial (RCT) of ITH versus delayed ITH to evaluate mental health effectiveness and ease of implementation.

DETAILED DESCRIPTION:
Background: Somalia has long been in a state of humanitarian crisis; trauma-related mental health needs are extremely high. Access to state-of-the-art mental health care is limited. Islamic Trauma Healing (ITH) is a manualized mosque-based, lay-led group intervention aimed at healing the individual and communal mental wounds of war and refugee trauma. The 6-session intervention combines Islamic principles with empirically-supported exposure and cognitive restructuring principles for posttraumatic stress disorder (PTSD). ITH reduces training time, uses a train the trainers (TTT) model, and relies on local partnerships embedded within the strong communal mosque infrastructure.

Methods: The investigators will conduct a hybrid effectiveness-implementation randomized control trial (RCT) in the Somaliland, with implementation in the cities of Hargeisa, Borama, and Burao. In this study, a lay-led, mosque-based intervention, Islamic Trauma Healing (ITH), to promote mental health and reconciliation will be examined in 200 participants, randomizing mosques to either immediate ITH or a delayed (waitlist; WL) ITH conditions. Participants will be assessed by assessors masked to condition at pre, 3 weeks, 6 weeks, and 3 month follow-up. Primary outcome will be assessor-rated posttraumatic stress symptoms (PTSD), with secondary outcomes of depression, somatic symptoms, and well-being. A TTT model will be tested, examining the implementation outcomes. Additional measures include potential mechanisms of change and economic evaluation.

Conclusion: This trial has the potential to provide effectiveness and implementation data for an empirically-based principle trauma healing program for the larger Islamic community that may not seek mental health care or does not have access to such care.

ELIGIBILITY:
Inclusion Criteria:

* Experienced a DSM-5 Criterion A trauma at least 12 weeks ago
* Report current re-experiencing or avoidance PTSD symptoms
* Islamic faith
* 18-70 years of age

Exclusion Criteria:

* Immediate suicide risk, with intent or plan
* Cannot understand consent/visible cognitive impairment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-05-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
PTSD Scale - Interview for the Diagnostic and Statistical Manual Version 5 | Change from pre to week 6 (immediate post intervention)
  PTSD Severity, higher score worse severity, 0 to 80

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 | Change from pre to week 6 (immediate post intervention)
  Depression Severity, higher score worse severity, 0 to 27
Somatic Symptoms Scale-8 | Change from pre to week 6 (immediate post intervention)
  Somatic Symptom Severity, higher score worse severity, 0 to 32
World Health Organization-5 Wellbeing Index | Change from pre to week 6 (immediate post intervention)
  Quality of Well-Being, higher score better well-being, 0 to 25

OTHER OUTCOMES:
Session Fidelity Checklist | ITH Session 1 through Session 6
  Session by session rating of adherence to the protocol, higher better, 0% to 100%, average items completed
Implementation Outcome Measure | Immediately post ITH intervention
  Acceptability, appropriateness, and feasibility, higher better, 1 to 5
Client Services Satisfaction Questionnaire | Immediately post ITH intervention
  Satisfaction with ITH, high score higher satisfaction, 5 to 20

CONTACTS AND LOCATIONS:
Overall Officials: Norah C Feeny, PhD, Principal Investigator — Case Western Reserve University; Jacob A Bentley, PhD, Principal Investigator — University of Washington; Lori A Zoellner, PhD, Principal Investigator — University of Washington
Locations (2):
- Somalia (2):
  - Somaliland Youth Development and Voluntary Organization, Burao
  - University of Burao, Burao

IPD SHARING:
Plan to Share IPD: Yes
Access to the data may be provided to qualified researchers engaging in independent scientific research on posttraumatic stress disorder. Data will be provided to the requesting party following review and approval of a research proposal, statistical analysis plan and execution of a Data Sharing Agreement. Data shared will be coded, with no personal health information included.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data request can be submitted starting 9 months after the article publication and data will be accessible for up to 24 months. Extensions will be considered on a case by case basis.
Access Criteria: Data will be provided to the requesting party following review and approval of a research proposal, statistical analysis plan, and execution of a Data Sharing Agreement.
  For more information or to submit a request, please contact zoellner@uw.edu.

REFERENCES:
- [Derived] Zoellner LA, Feeny NC, Angula DA, Aideed MH, Liban EN, Egeh MH, Awke AI, Ismail AS, Kunle MA, Ali E, Levin CE, Burant CJ, Bentley JA. Islamic trauma healing (ITH): A scalable, community-based program for trauma: Cluster randomized control trial design and method. Contemp Clin Trials Commun. 2023 Dec 10;37:101237. doi: 10.1016/j.conctc.2023.101237. eCollection 2024 Feb. PMID 38222876

DOCUMENTS (2):
  • Informed Consent Form: Main Study Consent English (2022-04-22): https://cdn.clinicaltrials.gov/large-docs/82/NCT05890482/ICF_000.pdf
  • Informed Consent Form: Group Leader Consent English (2022-04-22): https://cdn.clinicaltrials.gov/large-docs/82/NCT05890482/ICF_001.pdf